CLINICAL TRIAL: NCT00758745
Title: Randomized Contralateral Clinical Trial With Single-piece (SN60WF) vs. Three Piece (MA60AC) AcrySof Intraocular Lenses (IOLs) on Development of Posterior Chamber Opacification (PCO).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-06-03
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2011-07-28 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Cataract
Keywords: Cataract; Patients; bilateral; age related; undergoing; phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Model SN60WF (Active Comparator): Implantation with the AcrySof Model SN60WF Intraocular Lens (IOL)
  Interventions: Device: Model SN60WF
- Model MA60AC (Active Comparator): Implantation with the AcrySof Model MA60AC Intraocular Lens (IOL)
  Interventions: Device: Model MA60AC

INTERVENTIONS:
Device: Model SN60WF — Implantation with the AcrySof Model SN60WF Single-piece intraocular lens (IOL) following cataract removal.
  Arms: Model SN60WF
Device: Model MA60AC — Implantation with the AcrySof Model MA60AC multi-piece intraocular lens (IOL) following cataract surgery.
  Arms: Model MA60AC

SUMMARY:
Randomized contralateral clinical trial with single piece (Model SN60WF) vs. three piece (Model MA60AC) AcrySof Intraocular Lenses (IOLs) on development of Posterior Chamber Opacifiation (PCO).

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Clear cornea
* Pupil mydriasis ≥ 7mm
* In the bag Intraocular Lens (IOL)

Exclusion Criteria:

* Ocular pathology - uveitis, glaucoma, pseudoexfoliation syndrome (PEX), high myopia
* Previously operated eye
* Proliferative diabetic retinopathy
* Surgical complications - incomplete rhexis, post capsular rupture (PCR), zonular dialysis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Study Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Model SN60WF | Model MA60AC
Started | 81 | 81
Completed | 60 | 60
Not Completed | 21 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Model SN60WF | Model MA60AC | Total
Number analyzed (Participants) | 81 | 81 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 58 | 116
  >=65 years | 23 | 23 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 41 | 41 | 82

OUTCOME MEASURES:

1. Primary Outcome: Posterior Capsule Opacification (PCO)
Description: Development of PCO using the EPCO Score. The EPCO score incorporates planimetric & grading assessments. The density of the opacification behind the Intraocular Lens (IOL) is graded clinically as follows: 0=No detectable opacification; 1=Minimal detectable opacification; 2=mild detectable opacification; 3=moderate detectable opacification; 4=severe detectable opacification. The individual PCO score is calculated by multiplying the opacification grade by the fraction of capsule area involved behind the IOL optic. The selection process and grading of areas are subjective.
Time Frame: Up to 3 years
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Model SN60WF | Model MA60AC
Number analyzed (Participants) | 60 | 60
Units on a scale | 0.18 (0.41) | 0.15 (0.44)

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study.
Arm/Group | Model SN60WF | Model MA60AC
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/81
Other Adverse Events (participants affected / at risk) | 0/81 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data is held confidential and not be disclosed to a 3rd party without written consent from Alcon Laboratories for a period of 3 years.